CLINICAL TRIAL: NCT06644196
Title: Creation of a Database of Images of the Eye With the Holographic Doppler Laser
Acronym: IREDO
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SBN_2022_9
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Vessels of the Eye Fundus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Acquisition of images/videos of the bilateral fundus with the holographic doppler laser — Acquisition of images/videos of the bilateral fundus with the holographic Doppler laser

SUMMARY:
Many retinal pathologies are of vascular origin. In order to better understand their pathophysiology and make an accurate diagnosis, it is essential to visualise and quantify blood flow. The holographic Doppler laser (LDH) is a new medical device currently being developed by physics researchers at the Institut Langevin. The 1st prototype of this device is currently being used as part of research involving humans with minimal risks and constraints at the Hôpital National de la Vision des Quinze-Vingts (NCT04129021).

In order to better visualise, understand and quantify the vascular anomalies suspected in the fundus of patients undergoing ophthalmology treatment , we would like to acquire images/videos with a 2nd LDH prototype, within the ophthalmology clinical investigation platform at the Hôpital Fondation Adolphe de Rothschild.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Age ≥ 18 years
* Having received informed information about the study and having signed a consent to participate in the study
* Affiliated or beneficiary of social insurance

For participants with no known ocular pathology:

- No known ocular pathology other than a refractive disorder

For patients with optic nerve pathology:

- Patient undergoing ophthalmology consultation for optic nerve pathology in at least one eye (examples: glaucoma, optic neuritis, hereditary optic nerve diseases)

For patients with retinal and/or choroidal pathology:

- Patients undergoing ophthalmology consultations for retinal and/or choroidal pathology in at least one eye (examples: diabetic retinopathy, age-related macular degeneration).

For patients with retinal vascular pathology:

- Patient undergoing ophthalmology consultation for retinal vascular pathology in at least one eye (e.g. central retinal artery occlusion, central retinal vein occlusion, ocular ischemia syndrome).

Exclusion Criteria:

* Inability to maintain a stable sitting position
* Contraindications to holographic doppler laser :

  * implanted medical electronic device (pacemaker or other)
  * history of photosensitivity.
  * received photo-dynamic therapy (PDT) within the last 3 months.
  * viral conjunctivitis or any other infectious disease.
  * skin lesions on the neck or forehead, not allowing contact with a chin strap
  * patients at high risk of damage from optical radiation (e.g. aphakic patients, or patients with reduced sensitivity to light due to disease of the back of the eye).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from ophthalmology consultations , or for participants with no ocular pathology, from staff, patients followed for a non-ophthalmological pathology or patient companions.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-11-07 (Estimated); Study Completion 2026-11-07 (Estimated)

PRIMARY OUTCOMES:
Describe the usability of acquisitions (images/videos) of retinal and choroidal vascularization with holographic laser Doppler. | Day0
  Acquisitions (images/videos) will be considered usable if they allow :
  * (1) The ophthalmologist can visually distinguish arterial and venous vascular networks.
  * (2) The device measures arterial and venous blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Lejoyeux, Dr, Principal Investigator — Hôpital Fondation Adolphe de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschild, Paris, France